CLINICAL TRIAL: NCT03767218
Title: Initiation of Ovarian Stimulation With Recombinant-human FSH (Bemfola®) in the Late Follicular Phase, a Randomised Controlled Pilot Study.
Brief Title: Initiation of Ovarian Stimulation With Recombinant-human FSH (Bemfola®) in the Late Follicular Phase
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2.D12.Bemfola
Record Dates: First submitted 2018-05-17; First posted 2018-12-06 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2022-04

CONDITIONS: Infertility, Female
Keywords: Oocyte donor; Ovarian stimulation
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: Open label, phase 3 pilot randomized trial using a two-arm design with 1:1 allocation ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Late follicular phase stimulation with recombinant-human FSH (Experimental): Start of ovarian stimulation with recombinant-human FSH (Bemfola 225 IU daily) from the late follicular phase of the menstrual cycle onwards. Start of GnRH antagonist (ganirelix 0.25mg/day) when serum LH > 10 IU/L, till day of trigger.
  Interventions: Combination Product: Late follicular phase stimulation with recombinant-human FSH
- Early follicular phase stimulation with recombinant-human FSH (Active Comparator): Start of ovarian stimulation with recombinant-human FSH (Bemfola 225 IU daily) from day 2 of follicular phase onwards. Initiation of GnRH antagonist (ganirelix, 0.25mg/day) on stimulation day 6 till day of trigger.
  Interventions: Combination Product: Early follicular phase stimulation with recombinant-human FSH

INTERVENTIONS:
Combination Product: Late follicular phase stimulation with recombinant-human FSH — Start of ovarian stimulation with recombinant-human FSH (Bemfola 225 IU daily) from the late follicular phase of the menstrual cycle onwards. Start of GnRH antagonist (ganirelix 0.25mg/day) when serum LH > 10 IU/L, till day of trigger.
  Arms: Late follicular phase stimulation with recombinant-human FSH
Combination Product: Early follicular phase stimulation with recombinant-human FSH — Start of ovarian stimulation with recombinant-human FSH (Bemfola 225 IU daily) from day 2 of follicular phase onwards. Initiation of GnRH antagonist (ganirelix, 0.25mg/day) on stimulation day 6 till day of trigger.
  Arms: Early follicular phase stimulation with recombinant-human FSH

SUMMARY:
A randomised controlled open-label clinical trial to compare the outcome parameters after ovarian stimulation using recombinant-human FSH (follicle stimulating hormone), starting on day 2 of the cycle versus start in the late follicular phase of the cycle.

DETAILED DESCRIPTION:
Objective: To determine whether late follicular stimulation using recombinant-human FSH has comparable outcomes to treatment using recombinant-human FSH in early follicular phase in a flexible GnRH (Gonadotropin-releasing hormone) antagonist protocol, in oocyte donor patients.

Design: Open label, phase 3 randomized trial using a two-arm design with 1:1 allocation ratio

Patients: Oocyte donors (aged 18-36 years)

Intervention(s): Reference group: Start of ovarian stimulation with recombinant-human FSH (Bemfola 225 IU daily) from day 2 of follicular phase onwards. Initiation of GnRH antagonist (ganirelix, 0.25mg/day) on stimulation day 6 till day of trigger.

Investigational group: Start of ovarian stimulation with recombinant-human FSH (Bemfola 225 IU daily) from the late follicular phase of the menstrual cycle (evaluation trough ultrasound and hormonal assessment) onwards. Start of GnRH antagonist (ganirelix 0.25mg/day) when serum LH (Luteinizing Hormone) > 10 IU/L, till day of trigger.

Oocyte maturation trigger with GnRH agonist (0.2mg Gonapeptyl) in both groups.

ELIGIBILITY:
Inclusion Criteria:

* oocyte donor patients
* Age from 18 to 36 years
* BMI 19 to 35
* Regular menstrual cycle length i.e. 24-35 days

Exclusion Criteria:

* Patients with AMH <1.1 ng/ml and/or AFC<7
* Patients with FNPO (Follicle Number Per Ovary) ≥ 19 and/ord AMH >5ng/ml
* Endometriosis grade 3-4
* Oligo-amenorrhea
* Any untreated endocrine abnormality

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
total amount of COC (cumulus-oocyte-complex) | at oocyte aspiration

SECONDARY OUTCOMES:
Endocrine profile | on menstrual cycle day 2 9, (extra days as per site protocol) and day of oocyte maturation trigger in reference group. On menstrual cycle day 2 and 12, (extra days as per site protocol) and day of oocyte maturation trigger in investigational group
  LH (Luteinising hormone) level
Endocrine profile | on menstrual cycle day 2 and 9, (extra days as per site protocol) and day of oocyte maturation trigger in reference group. On menstrual cycle day 2 and 12, (extra days as per site protocol) and day of oocyte maturation trigger in investigational group
  FSH level
Endocrine profile | on menstrual cycle day 2 and 9, (extra days as per site protocol) and day of oocyte maturation trigger in reference group. On menstrual cycle day 2 and 12, (extra days as per site protocol) and day of oocyte maturation trigger in investigational group
  Progesterone level
Endocrine profile | on menstrual cycle day 2 and 9, (extra days as per site protocol) and day of oocyte maturation trigger in reference group. On menstrual cycle day 2 and 12, (extra days as per site protocol) and day of oocyte maturation trigger in investigational group
  Estradiol level
Consumption of gonadotrophins | during the ovarian stimulation
  totaal amount of IU (international units) used
Number of days needed for ovarian stimulation | during the ovarian stimulation
Days of GnRH antagonist use | during the ovarian stimulation
Total number of mature oocytes | at day of oocyte aspiration
Total medication cost | during the ovarian stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR